CLINICAL TRIAL: NCT04425317
Title: Detection of SARS-CoV-2 in Follicular Fluid and Cumu-lus-oocyte-complexes From COVID-19 Patients During Controlled Ovarian Stimulation for ICSI Treatment
Brief Title: Detection of SARS-CoV-2 in Follicular Fluid and Cumulus-oocyte-complexes in COVID-19 Patients
Acronym: COVID_OFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CRG UZ Brussel (Other)
Responsible Party: Principal Investigator, Liese Boudry, MD, CRG UZ Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVIDOFF001
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Infertility; COVID; IVF
MeSH Terms: conditions — Infertility | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic arm (Other): Blood sample and endometrial biopsy Collection of follicular fluid, immature oocytes and cumulus cells
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample and endometrial biopsy on the moment of oocyte retrieval
  Other Names: Endometrial biopsy

SUMMARY:
Recently, the world was shaken awake by a pandemic caused by a novel coronavirus SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2). In most nations drastic isolation measures were taken to minimize the further spread of the Coronavirus Disease 2019 (COVID-19). Being the first pandemic sparked by a Coronavirus, little was known on COVID-19 and its implications on general health. Our understanding on the virus and its potential effects on health is growing. In Belgium, the situation is stabilizing, and doctors and healthcare workers are slowly recommencing routine work and consultations. As also fertility treatments were abruptly interrupted, many patients are in need to resume their treatment. The limited evidence of SARS-CoV-2 on pregnancy seems to be rather satisfying1, but practically nothing is known about the possible impact of an active SARS-CoV-2 infection on female gametes. Viral transmission occurs predominantly through respiratory droplets, but transmission to gametes cannot be ruled out.

Since the onset of the pandemic, knowledge about the molecular details of SARS-CoV-2 infection rapidly grew. Coronaviruses are enveloped RNA viruses. For a virus to deliver their genome into the host cell, attachment and entrance into that cell is a crucial step. The coronavirus surface protein spike (S) mediates entry into target cells by binding to a cellular receptor and subsequent fusing of the viral envelope with a host cell membrane. The SARS-CoV-2-S protein (SARS-S) utilizes angiotensin-converting enzyme 2 (ACE2) as a receptor for host cell entry. Host proteases such as transmembrane serine protease 2 (TMPRSS2) are then needed to cleave the viral S protein, allow-ing permanent fusion of the viral and host cell membranes2. Expression of ACE2 and TMPRSS2 has been shown in testicular, uterine and placental cells. Based on available transcriptomic data, co-expression of ACE2 and TMPRSS2 is also seen on oocyte level, but the possible impact on reproduction is unknown. The BSG (basigin or CD147), a receptor on host cells, was also identified as a possible route for viral invasion.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Undergoing IVF/ICSI treatment
* Planned for an oocyte retrieval
* PCR positive of SARS-CoV-2 or high suspicion for COVID 19 based on CT scan
* Signed informed consent

Exclusion Criteria:

* None

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of SARS-CoV-2 in follicular fluid, cumulus cells, immature oocytes and endometrium | 1 day
  Identification of viral RNA in cumulus-oocyte-complexes, exclusively looking at the material that is considered waste material in a normal oocyte retrieval

SECONDARY OUTCOMES:
Presence of ACE2, TMPRSS and BSG receptors in cumulus cells, immature oocytes and endometrium | 1 day
  Presence of receptors, identified as possible steps in the entry pathway for SARS-CoV-2

CONTACTS AND LOCATIONS:
Locations (1):
- Uz Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hou R, Huang R, Zhou Y, Lin D, Xu J, Yang L, Wei X, Xie Z, Zhou Q. Single-cell profiling of the microenvironment in decidual tissue from women with missed abortions. Fertil Steril. 2023 Mar;119(3):492-503. doi: 10.1016/j.fertnstert.2022.12.016. Epub 2022 Dec 15. PMID 36528108
- [Derived] Boudry L, Essahib W, Mateizel I, Van de Velde H, De Geyter D, Pierard D, Waelput W, Uvin V, Tournaye H, De Vos M, De Brucker M. Undetectable viral RNA in follicular fluid, cumulus cells, and endometrial tissue samples in SARS-CoV-2-positive women. Fertil Steril. 2022 Apr;117(4):771-780. doi: 10.1016/j.fertnstert.2021.12.032. Epub 2022 Jan 1. PMID 35272846